CLINICAL TRIAL: NCT00738166
Title: Content, Bioavailability and Health Effects of Trace Elements and Bioactive Components in Organic Agricultural Systems
Acronym: OrgTrace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H-C-2007-0078; M194
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: diet, organic, health; healthy people
MeSH Terms: interventions — Diet; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- II (Experimental): organic animal manure
  Interventions: Other: Organic or conventional diet; Other: Diet (organic or conventional)
- III (Active Comparator): conventional
  Interventions: Other: Organic or conventional diet; Other: Diet (organic or conventional)
- I (Experimental): organic green manure
  Interventions: Other: Organic or conventional diet; Other: Diet (organic or conventional)

INTERVENTIONS:
Other: Organic or conventional diet — 12 days on fully controlled organic 1 diet, organic 2 diet and conventional diet
Other: Diet (organic or conventional) — organic or conventional diet

SUMMARY:
Trace elements, bioactive secondary metabolites and vitamins are among the most important quality parameters in plants. Yet, very little information is available on their content, bioavailability and health effects of organically grown plant food products. The main objective of the project is to study the impact of different agricultural management practises relevant for organic farming on the ability of cereal and vegetable crops to absorb trace elements from the soil and to synthesise bioactive compounds (secondary metabolites, antioxidant vitamins and phytates) with health promoting effects. Field experiments with a rigidly controlled design will be implemented together with state-of-the-art analytical techniques allowing solid conclusions to be drawn on the variability and optimum levels of bioactive compounds. The multitude of analytical data from plant and soil samples will be analysed by multivariate statistical methods in order to reveal differences between the cultivation systems used. Finally, the relationship between bioavailability of the nutrients studied and the elemental fingerprint of plants will be extracted by the statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-45 years
* BMI 20-30 kg/m2
* Non-vegetarian

Exclusion Criteria:

* Physical activity > 10 h/week
* Intake of dietary supplements
* Regular use of drugs
* Chronic diseases
* Smoking
* Excessive intake of alcohol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability of trace elements and secondary metabolites | 3 x 12 days

SECONDARY OUTCOMES:
Health factors | 3 x 12 days

OTHER OUTCOMES:
miRNA | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- IHE-LIFE, Frederiksberg, Denmark